CLINICAL TRIAL: NCT04382170
Title: Dexmedetomidine Sublingual Film for the Management of Agitation in Delirium: Safety and Preliminary Efficacy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study sponsor decided not to perform this study.
Sponsor: Jeff C. Huffman, MD (Other)
Collaborators: BioXcel Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Jeff C. Huffman, MD, Director of the Cardiac Psychiatry Research Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P002353
Record Dates: First submitted 2020-04-25; First posted 2020-05-11 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Delirium
Keywords: agitation; delirium; dexmedetomidine
MeSH Terms: conditions — Delirium; Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, controlled, 2-arm, double-blinded trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20 mcg (Active Comparator): Participants randomized to the 20mcg group will receive 20mcg of dexmedetomidine sublingual film every 30 minutes, if they continue to have agitation and do not meet any cardiovascular stopping criteria. The maximum dosing for this arm is 80mcg.
  Interventions: Drug: Dexmedetomidine sublingual film
- 60 mcg (Experimental): Participants randomized to the 60mcg group will receive 60mcg of dexmedetomidine sublingual film every 30 minutes, if they continue to have agitation and do not meet any cardiovascular stopping criteria. The maximum dosing for this arm is 240mcg.
  Interventions: Drug: Dexmedetomidine sublingual film

INTERVENTIONS:
Drug: Dexmedetomidine sublingual film — Dexmedetomidine sublingual film for the management of agitation in hospitalized patients with delirium.
  Other Names: Precedex

SUMMARY:
The investigator will examine the safety, tolerability, optimal dose, and preliminary efficacy of dexmedetomidine sublingual film in a randomized, double-blind, controlled trial in 40 hospitalized patients with hyperactive delirium (i.e., delirium with agitation) in the Intensive Care Unit (ICU) setting.

Specific Aim #1 (safety and tolerability): To examine the incidence of cardiovascular and other side effects following the administration of dexmedetomidine sublingual film in patients hospitalized in the ICU with delirium and agitation in a randomized, double-blind trial (total N=80 patients with delirium [with or without agitation], with a goal of administering dexmedetomidine to at least 40 participants with agitation).

Hypothesis: Dexmedetomidine sublingual film will be associated with hypotension and/or bradycardia requiring clinical intervention in ≤ 20% (8 of 40) participants. Dexmedetomidine will not be associated with QTc prolongation or non-cardiac adverse events.

Specific Aim #2 (preliminary efficacy): To examine the impact of dexmedetomidine sublingual film on agitation and delirium severity.

Hypothesis: Dexmedetomidine will lead to reductions in agitation and delirium severity during the follow-up period (co-primary endpoints = 1 and 2 hours post-administration).

Specific Aim #3 (optimal dosing): To identify the minimum dose that is effective at reducing agitation and delirium severity without causing significant side effects.

Hypothesis: Participants receiving doses of 60 mcg of dexmedetomidine will have a faster time to a reduction in agitation and greater reductions in delirium severity than participants receiving 20 mcg of dexmedetomidine.

DETAILED DESCRIPTION:
Study Intervention

Participants will be randomized to receive either 20 mcg or 60 mcg of dexmedetomidine sublingually. Participants will receive repeat dosing every 30 minutes for up to three additional doses, leading to maximum doses of 80 mcg and 240 mcg, respectively. Both investigators and clinicians will be blind to the participant's group, with only the study pharmacist aware of the dose of medication on the films.

Baseline monitoring: Following enrollment, the study team will record baseline measures of heart rate, blood pressure, and oxygen saturation. An electrocardiogram (ECG) will be performed, and agitation and delirium severity will be measured.

Medication administration: Dexmedetomidine sublingual film will be administered by the study physician or study nurse as per the manufacturer's instructions. Dexmedetomidine administration will be repeated every 30 minutes if the participant continues to have agitation and does not meet any cardiovascular stopping criteria.

Monitoring for side effects: Heart rate, blood pressure, oxygen saturation, use of supplemental oxygen, and use of pressors will be monitored continuously and recorded every 30 minutes for the 6 hours following the initial medication administration (baseline; Time 0). An ECG will be performed at 1.5, 3, 4.5, and 6 hours, and QTc will be calculated using the Fridericia formula. Study staff will also monitor the participant and speak with nursing staff at 6 hours to assess for any other side effects/complaints the patient may have had during the time since medication administration.

Monitoring of agitation and delirium severity: Agitation will be measured every 30 minutes and delirium severity at hours 1, 2, 3, 4, and 6.

Study Endpoints

Safety and Tolerability (Aim #1) The investigators will examine changes in heart rate, blood pressure, oxygen saturation, and QTc interval from baseline to the follow-up timepoints, as well as the incidence of self-reported and clinician-reported side effects during the 6-hour post-medication interval. They also will record the total dosage of medication each participant received and examine whether medication dose was associated with the incidence of side effects.

Preliminary Efficacy (Aim #2) The investigators will assess changes in agitation and delirium from baseline to the follow-up timepoints. One and two hours following medication administration will be considered the co-primary timepoints for these efficacy measures. They also will record the total dosage of medication each participant received and examine whether medication dose was associated with a reduction in agitation and delirium severity.

Minimum Dose of Administration (Aim #3) The investigators will measure the amount of time from the initial dexmedetomidine administration until agitation resolves. Then, they will compare between-group differences in time to agitation resolution, changes in agitation and delirium severity, and the incidence of side effects. The optimal dose will be chosen based on the dose that leads to the quickest resolution of agitation without leading to clinically significant side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized on a medical or surgical intensive care unit at MGH
* Diagnosis of delirium, assessed according to DSM-5 criteria (DSM-5)
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, at screening
* Weight at least 60 kg (132 pounds), at screening
* In the opinion of the study and clinical teams, sufficiently physically healthy to receive dexmedetomidine sublingual film

Exclusion Criteria:

* Per medical record or team report, diagnoses of:

  * Dementia
  * Significant traumatic brain injury
  * History of stroke, with persistent neurologic deficits
* Presence of any of the following cardiovascular comorbidities

  * Sick sinus syndrome
  * A resting heart rate of < 55 beats per minutes or systolic blood pressure (BP) <100 mmHg or >160 mmHg or diastolic BP <70 mmHg or ˃ 95 mmHg at enrollment and prior to dosing.
  * Evidence of cardiac ischemia on a 12-lead electrocardiogram (ECG)
  * Corrected QT interval of > 450 msec
  * Presence of a permanent pacemaker device
* Per medical record (notes, current medications, flowsheets):

  * Second degree (or greater) Atrioventricular (AV) block without a pacemaker
  * Known allergy or adverse reaction to dexmedetomidine
  * Current use of dexmedetomidine
* Inability to take sublingual dexmedetomidine due to severe agitation, neurological impairment, nil per os (NPO) status, or other cause.
* Hepatic impairment (liver function tests > 3 times the upper limit of normal)
* Severe renal impairment (glomerular filtration rate (GFR) < 30 ml/min or on dialysis)
* Weight < 60 kg
* Pregnancy (in women; tested with serum or urine human chorionic gonadotropin [hCG])
* Non-fluency in English
* Prior enrollment in the study, with receipt of study medication, during the current or a previous hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate | Baseline, Medication Administration (Hour 0), Hour 0.5, Hour 1, Hour 1.5, Hour 2, Hour 2.5, Hour 3, Hour 3.5, Hour 4, Hour 4.5, Hour 5, Hour 5.5, Hour 6
  Heart rate will be assessed participant's flowsheet or using the telemetry monitor for the 6 hours following the initial medication administration.
Change in Blood Pressure | Baseline, Medication Administration (Hour 0), Hour 0.5, Hour 1, Hour 1.5, Hour 2, Hour 2.5, Hour 3, Hour 3.5, Hour 4, Hour 4.5, Hour 5, Hour 5.5, Hour 6
  Blood pressure will be assessed participant's flowsheet or using the telemetry monitor/automated blood pressure cuff for the 6 hours following the initial medication administration.
Change in Oxygen Saturation | Baseline, Medication Administration (Hour 0), Hour 0.5, Hour 1, Hour 1.5, Hour 2, Hour 2.5, Hour 3, Hour 3.5, Hour 4, Hour 4.5, Hour 5, Hour 5.5, Hour 6
  Oxygen saturation will be assessed participant's Epic flowsheet or using the telemetry monitor/pulse oximter for the 6 hours following the initial medication administration.
Change in QTc Interval | Baseline, Hour 1.5, Hour 3, Hour 4.5, Hour 6
  An ECG will be performed intermittently over the 6 hour monitoring period, and QTc will be calculated using the Fridericia formula.
Self-reported Side Effects | Hour 6
  Incidence of side effects reported for dexmedetomidine in post-marketing surveillance

SECONDARY OUTCOMES:
Change in Agitation | Baseline, Hour 0.5, Hour 1, Hour 1.5, Hour 2, Hour 2.5, Hour 3, Hour 3.5, Hour 4, Hour 4.5, Hour 6
  Agitation will be measured by the Richmond Agitation-Sedation Scale (RASS). RASS is a 10-point scale ranging from -5 to +4, with a more positive score indicating increased agitation.
Change in Delirium Severity | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6
  Delirium severity will be measured by the Delirium Rating Scale-revised-98 (DRS-R-98). The maximum possible score for severity items is 39, while the maximum total score is 46. Higher scores indicate more severe delirium; score of 0 indicates no delirium.
Time to resolution of agitation | Hour 6
  Amount of time from the initial dexmedetomidine administration until agitation resolves measured by RASS score < 1

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No